CLINICAL TRIAL: NCT06747026
Title: Real-world Survival Outcomes and the Evaluation of Optimal Strategies for Immuno-Radiotherapy in Advanced Non-Small-Cell Lung Cancer: a Territory-wide Study (OCEANUS Study)
Brief Title: Real-World Immuno-Radiotherapy for Advanced NSCLC
Acronym: OCEANUS
Status: Completed | Type: Observational
Sponsor: Fengming Kong (Other)
Responsible Party: Sponsor-Investigator, Fengming Kong, professor, The University of Hong Kong-Shenzhen Hospital
Organization: The University of Hong Kong-Shenzhen Hospital (Other)
Other Study IDs: Immuno-radiotherapy in NSCLC; UW 23-623 (Registry Identifier: HKU/HA HKW IRB)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer Non-Small Cell Cancer (NSCLC)
Keywords: advanced NSCLC; ICIs; radiotherapy; iRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- initial iRT for locally advanced NSCLC: For unresectable locally advanced NSCLC: definitive thoracic radiotherapy must have been administered as the initial treatment, with immunotherapy initiated within 90 days after RT (Sequential iRT) or concurrently with RT (Concurrent iRT).
  Interventions: Drug: initial Sequential iRT; Drug: initial Concurrent iRT
- initial iRT for de novo metastatic NSCLC: For de novo metastatic NSCLC: radiotherapy targeting the primary lung tumor or metastatic lesions must have been administered as the initial treatment, with immunotherapy initiated within 90 days after RT (Sequential iRT) or concurrently with RT (Concurrent iRT).
  Interventions: Drug: initial Sequential iRT; Drug: initial Concurrent iRT
- Salvage iRT in post-treatment progressive NSCLC: For post-treatment progressive NSCLC: salvage radiotherapy must have been performed during immunotherapy or within 90 days after the cessation of immunotherapy (RT after discontinuation of ICI) , or concurrently with RT (RT with maintenance of ICI).
  Interventions: Drug: RT with maintenance of ICI; Drug: RT after discontinuation of ICI

INTERVENTIONS:
Drug: initial Sequential iRT — For unresectable locally advanced NSCLC, definitive thoracic radiotherapy must have been administered as the initial treatment, with immunotherapy initiated within 90 days after RT.
  For de novo metastatic NSCLC, radiotherapy targeting the primary lung tumor or metastatic lesions must have been administered as the initial treatment, with immunotherapy initiated within 90 days.
  Groups: initial iRT for de novo metastatic NSCLC; initial iRT for locally advanced NSCLC
Drug: initial Concurrent iRT — For unresectable locally advanced NSCLC, definitive thoracic radiotherapy must have been administered as the initial treatment, with immunotherapy concurrently with RT.
  For de novo metastatic NSCLC, radiotherapy targeting the primary lung tumor or metastatic lesions must have been administered as the initial treatment, with immunotherapy concurrently with RT.
  Groups: initial iRT for de novo metastatic NSCLC; initial iRT for locally advanced NSCLC
Drug: RT with maintenance of ICI — For post-treatment progressive NSCLC, salvage radiotherapy performed during immunotherapy.
  Groups: Salvage iRT in post-treatment progressive NSCLC
Drug: RT after discontinuation of ICI — For post-treatment progressive NSCLC, salvage radiotherapy performed during within 90 days after the cessation of immunotherapy.
  Groups: Salvage iRT in post-treatment progressive NSCLC

SUMMARY:
The optimal combination strategy for radiotherapy combined with immunotherapy (iRT) in advanced non-small-cell lung cancer (NSCLC) remains unclear, and there is a lack of real-world data to validate its efficacy. The objective of this study is to confirm the survival benefits of iRT in advanced NSCLC and to identify the optimal combination strategy for its use.

DETAILED DESCRIPTION:
The PACIFIC study has established radiotherapy combined with immune checkpoint inhibitors (iRT) as the primary treatment modality for unresectable, locally advanced non-small-cell lung cancer (NSCLC). Simultaneously, the KEYNOTE-001 study provided evidence supporting the efficacy of iRT in patients with metastatic and progressive NSCLC. However, most available evidence comes from interventional clinical trials, where participants are rigorously selected and required to adhere strictly to protocol-defined interventions. This creates a significant gap in real-world data, which is essential to further validate the survival benefits of iRT in advanced NSCLC. Furthermore, clinical trials evaluating concurrent iRT in NSCLC have largely yielded negative or inconclusive results, highlighting the need for clarity on the optimal combination strategy for iRT.

To address these gaps, researchers will conduct a territory-wide real-world cohort study. The objective of this study is to validate the survival benefits of iRT in patients with advanced NSCLC and to identify the optimal sequential strategy for iRT.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC patients who received immunotherapy between 2015 and 2021
* For unresectable locally advanced NSCLC: definitive thoracic radiotherapy must have been administered as the initial treatment, with immunotherapy initiated within 90 days after RT or concurrently with RT
* For de novo metastatic NSCLC: radiotherapy targeting the primary lung tumor or metastatic lesions must have been administered as the initial treatment, with immunotherapy initiated within 90 days after RT or concurrently with RT
* For post-treatment progressive NSCLC: salvage radiotherapy must have been performed during immunotherapy or within 90 days after the cessation of immunotherapy
* Age >= 18 years old

Exclusion Criteria:

* Patients with multiple primary cancers or a pathological diagnosis of small cell lung cancer
* Patients who did not receive radiotherapy or who did not undergo radiotherapy within 90 days before or after immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced NSCLC patients undergo immunotherapy combined with radiotherapy.
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
OS (overall survival) | From the initiation date of iRT to the date of death from any cause, with a follow-up period of up to approximately 5 years.
  OS is defined as the time from the initiation of iRT until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, HongKong, Hong Kong

IPD SHARING:
Plan to Share IPD: No